CLINICAL TRIAL: NCT02470754
Title: Clinical Pharmacology of Electronic Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Roswell Park Cancer Institute (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15635; R01DA039264 (NIH); NCI-2018-02897 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2015-04-30; First posted 2015-06-12 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EC Block1/TC Block 2 (Active Comparator): Participants will be randomized into one of two groups. In this group, participants will be assigned to Electronic Cigarettes only for Study Block #1, then crossover to Tobacco Cigarettes only for Study Block #2.
  Interventions: Device: Tobacco Cigarette; Device: Electronic Cigarette
- TC Block 1/EC Block 2 (Active Comparator): Participants will be randomized into one of two groups. In this group, participants will be assigned to Tobacco Cigarettes only for Study Block #1, then crossover to Electronic Cigarettes only for Study Block #2.
  Interventions: Device: Tobacco Cigarette; Device: Electronic Cigarette

INTERVENTIONS:
Device: Tobacco Cigarette — Usual brand tobacco cigarette smoked by study participant.
  Other Names: TC, Cigarette
Device: Electronic Cigarette — Usual brand electronic cigarettes smoked by study participant.
  Other Names: EC, E-cig, E-cigarette

SUMMARY:
The purpose of this study is to learn more about nicotine exposure and the safety of electronic cigarettes (EC). It will focus on the areas that are thought to most closely relate to the addictive potential of EC, namely: (1) EC as nicotine delivery devices, covering issues of nicotine intake and pharmacokinetics, temporal patterns of use and titration of nicotine; and (2) subjective effects of EC use, including relationship of use to reward, withdrawal and craving.

DETAILED DESCRIPTION:
Electronic cigarettes (EC) are nicotine delivery devices that generate a nicotine-containing aerosol which is inhaled by the user. EC are perceived by users to be useful in helping quitting smoking of conventional tobacco cigarettes (TC) as well as having a presumed lower risk of adverse health effects compared to TC, the potential for use in public places, reduced cost, and lack of the noxious clinging odors associated with TC use. Many believe that electronic cigarette (EC) function as nicotine delivery devices in the same way as tobacco cigarettes (TC), and that EC will prove to be just as addictive as TC, but this may not be the case because of fundamental differences in the design and method of use of these products. Investigators hypothesize that systemic nicotine exposure will be lower with EC compared to TC; that despite lower nicotine intake EC users will experience similar reward and no greater withdrawal symptoms or craving compared to TC; and that dual EC/ TC users will not titrate their daily intake of nicotine in the same way that TC smokers of high- vs low-yield nicotine TC do.

Investigators specifically focus on the areas that are thought to most closely relate to the addictive potential of EC, namely: (1) EC as nicotine delivery devices, covering issues of nicotine intake and pharmacokinetics, temporal patterns of use and titration of nicotine; and (2) subjective effects of EC use, including relationship of use to reward, withdrawal and craving. The investigators will also examine aspects of safety of EC use (by assessment of cardiovascular and hormonal effects of use and of biomarkers of exposure to potentially toxic constituents) and explore the identification and validation of biomarkers that may be useful in distinguishing EC from TC use. Study subjects will be dual users of TC and EC so that the investigators may compare both modalities of use in experienced users in a within-subject design.

The study will consist of two 1-week blocks (EC-only or TC-only conditions) with 4 days of outpatient ad libitum product use followed by 3 days in a clinical research ward to include a single-use pharmacokinetic study, monitoring of product use, subjective assessments, blood and urine collections to assess biomarkers, and a 24-hour period of cardiovascular monitoring. Two additional days at the end of the 2nd block will assess similar measurements during a period of nicotine-product abstention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of medical history and limited physical examination as described below:

  * Heart rate < 105 BPM*
  * Systolic Blood Pressure < 160 and > 90*
  * Diastolic Blood Pressure < 100 and > 50*
  * Body Mass Index ≤ 38.0 *Considered out of range if both machine and manual readings are above/below these thresholds.
* Current regular "dual" user of both EC and conventional TC
* EC device is one of the most popular 1st, 2nd or 3rd generation brands (with the exception of rebuildable atomizers) as determined at time of study commencement
* Carbon monoxide ≥ 5 ppm or per discretion of Principal Investigator
* Saliva cotinine ≥50 ng/ml or urine cotinine
* Age: ≥ 21 years

Exclusion Criteria:

* Current regular use of selected psychiatric medications
* Current regular use of cardiovascular medications for cardiovascular conditions including hypertension (Example: beta and alpha-blockers)
* Current regular use of medications inducers of nicotine metabolizing enzymes CYP2A6 (Example: rifampicin, dexamethasone, phenobarbital, and other anticonvulsant drugs).
* Use of other tobacco products
* Pregnancy or breastfeeding (by history and pregnancy test)
* Concurrent use of nicotine-containing medications
* Drug/Alcohol Dependence
* Positive toxicology test at the screening visit (THC okay)
* Concurrent participation in another clinical trial
* Inability to communicate in English
* Planning to quit smoking within the next 60 days

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-07-23 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal L Benowitz, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco General Hospital (SFGH), San Francisco, California
  - University of California, San Francisco (UCSF), San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benowitz NL, St Helen G, Nardone N, Addo N, Zhang JJ, Harvanko AM, Calfee CS, Jacob P 3rd. Twenty-Four-Hour Cardiovascular Effects of Electronic Cigarettes Compared With Cigarette Smoking in Dual Users. J Am Heart Assoc. 2020 Dec;9(23):e017317. doi: 10.1161/JAHA.120.017317. Epub 2020 Nov 19. PMID 33208019

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EC Block1/TC Block 2 | TC Block 1/EC Block 2
Started | 19 | 19
Completed | 17 | 19
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Completers: all completed
Arm/Group | Completers
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black | 3
  Latino | 4
  White | 22
  Mixed | 5
Region of Enrollment [Number; unit: participants]
  United States | 36
Cigarettes per day [Mean (Standard Deviation); unit: Cigarettes per day] | 12.9 (6.4)
Days of EC use in past 30 [Mean (Standard Deviation); unit: Days] | 22.6 (7.3)
EC times per day [Mean (Standard Deviation); unit: Sessions per day] | 8.1 (7.2)
E-Cigarette Use index [Mean (Standard Deviation); unit: units on a scale] — E-Cigarette (EC) Use Index calculated as a function of (# of E-Cigarette Sessions Per Day) x E-Cigarette use days per Month) /30. Ranges from [0 to Infinity]. With lower values indicating minimal e-cigarette use and higher values indicating heavy E-Cigarette Use.
  units on a scale | 6.5 (6.5)
EC to TC use ratio [Mean (Standard Deviation); unit: ratio] | 0.57 (0.56)
Fagerstrom Test for Cigarette Dependence [Mean (Standard Deviation); unit: units on a scale] — The Fagerström Test for Nicotine Dependence is a standard instrument for assessing the intensity of physical addiction to nicotine.It contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence.Questionnaire scored 0-10 points with Total Score equal to the sum of all points.A patient who scores between 1 and 2 Test is classified as having a low dependence on nicotine. A patient who scores 5 and over would be considered highly dependent on nicotine.
  units on a scale | 4.4 (2.0)
Time to first cigarette [Count of Participants; unit: Participants] — Participant response to "How soon after you wake up do you usually have your first cigarette?" at baseline visit
  Participants
    ≤ 5 min | 6
    5-30 min | 21
    30-60 min | 8
    >60 min | 1
Time to first vape [Count of Participants; unit: Participants] — Participant response to "How soon after you wake up do you usually first use your e-cigarette?" at baseline visit
  Participants
    ≤ 5 min | 1
    5-30 min | 12
    30-60 min | 4
    > 60 min | 19
Salivary cotinine [Mean (Standard Deviation); unit: ng/mL] | 189 (92.8)
EC type [Count of Participants; unit: Participants]
  Cig-a-like | 12
  Fixed-power | 15
  Variable-power | 6
  Pod | 3
Flavor category [Count of Participants; unit: Participants]
  Dessert/candy | 8
  Fruit | 5
  Menthol | 5
  Tobacco | 18

OUTCOME MEASURES:

1. Primary Outcome: Standardized Session: Mean CMax
Description: Maximum Plasma Nicotine Concentration (Cmax) (ng/mL)
Time Frame: Inpatient Day 1, Up to 4 Hours post Nicotine Administration
Population: Pod users excluded
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Electronic Cigarette: EC ARM
- Combustible Cigarette: TC ARM
Arm/Group | Electronic Cigarette | Combustible Cigarette
Number analyzed (Participants) | 33 | 33
ng/mL | 6.1 (5.5) | 20.2 (11.1)

2. Primary Outcome: Standardized Session: Mean TMax
Description: Time (min) when Max Plasma Nicotine Concentration was achieved
Time Frame: Inpatient Day 1, Up to 4 Hours post Session
Population: Pod users excluded
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Electronic Cigarette | Combustible Cigarette
Number analyzed (Participants) | 33 | 33
minutes | 6.5 (5.4) | 2.7 (2.4)

3. Primary Outcome: Standardized Session: AUC 0-240
Description: Plasma Nicotine area-under-the curve from 0 to 4 Hours (min*ng/ml)
Time Frame: Inpatient Day 1, Up to 4 Hours post Session
Population: Pod users excluded
Measure: Mean (Standard Deviation); unit: min*ng/ml
Arm/Group | Electronic Cigarette | Combustible Cigarette
Number analyzed (Participants) | 33 | 33
min*ng/ml | 550 (438) | 1368 (665)

4. Primary Outcome: PK-estimated Nicotine Dose
Description: Estimated in dose received (in milligrams) during the Standardized Session.
Time Frame: Inpatient Day 1, Up to 4 Hours post Session
Population: Pod Users Excluded
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Electronic Cigarette | Combustible Cigarette
Number analyzed (Participants) | 33 | 33
mg | 0.9 (0.7) | 2.2 (1.2)

5. Secondary Outcome: Standardized Session: QSU Factor 1 (Vaping)
Description: Questionnaire for Smoking Urges Brief modified for e-cigarettes to measure urge to vape.Two factor scores and a total score were derived. Factor 1 represents the desire and intention to smoke with smoking perceived as rewarding, while Factor 2 represents an anticipation of relief from negative effect with an urgent desire to smoke.Scores range from 5 to 35 with higher scores indicating a higher level of craving.
Time Frame: Inpatient Day 1, Up to 4 Hours post Session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electronic Cigarette | Combustible Cigarette
Number analyzed (Participants) | 33 | 33
score on a scale | 23.9 (8.6) | 20.7 (10.0)

6. Secondary Outcome: Standardized Session: Positive and Negative Affect Score (Negative Affect)
Description: The PANAS Scale or Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire. PANAS, (Sandín et al., 1999; Watson, Clark & Tellegen, 1988).This instrument is composed of 20 items: 10 items measuring positive affective states and 10 items measuring negative affect states.This subscale measures a person's negative emotions. Scores range from 10- 50 with higher scores indicating stronger negative feelings.
Time Frame: Inpatient Day 1, Up to 4 Hours post Session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electronic Cigarette | Combustible Cigarette
Number analyzed (Participants) | 33 | 33
score on a scale | 14.3 (5.6) | 14.0 (5.0)

7. Secondary Outcome: Standardized Session: Minnesota Nicotine Withdrawal Scale
Description: Minnesota Nicotine Withdrawal Scale (MNWS) is a Self-Report Scale for measuring the severity of nicotine withdrawal symptoms.The possible range of scores for the 12-Item MNWS is between 0 and 48 with higher scores indicated greater withdrawal symptom severity.
Time Frame: Inpatient Day 1, Up to 4 Hours post Session
Population: Pod Users Excluded
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electronic Cigarette | Combustible Cigarette
Number analyzed (Participants) | 33 | 33
score on a scale | 10.8 (7.9) | 9.6 (7.4)

8. Secondary Outcome: Standardized Session: QSU Factor 2 (Vaping)
Description: Questionnaire for Smoking Urges Brief modified for e-cigarettes to measure urge to vape.Two factor scores and a total score were derived. Factor 1 represents the desire and intention to smoke with smoking perceived as rewarding, while Factor 2 represents an anticipation of relief from negative effect with an urgent desire to smoke. Scores range from 5 to 35 with higher scores indicating a higher level of craving.
Time Frame: Inpatient Day 1, Up to 4 Hours post Session
Population: Pod Users Excluded
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electronic Cigarette | Combustible Cigarette
Number analyzed (Participants) | 33 | 33
score on a scale | 14.9 (6.8) | 13.0 (7.0)

9. Secondary Outcome: Standardized Session: QSU Factor 1 (Smoking)
Description: Questionnaire for Smoking Urges Brief measures urge to smoke.Two factor scores and a total score were derived. Factor 1 represents the desire and intention to smoke with smoking perceived as rewarding, while Factor 2 represents an anticipation of relief from negative effect with an urgent desire to smoke. Scores range from 5 to 35 with higher scores indicating a higher level of craving.
Time Frame: Inpatient Day 1, Up to 4 Hours post Session
Population: Pod Users Excluded
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electronic Cigarette | Combustible Cigarette
Number analyzed (Participants) | 33 | 33
score on a scale | 22.9 (9.8) | 24.2 (9.9)

10. Secondary Outcome: Standardized Session: QSU Factor 2 (Smoking)
Description: as for outcome 9
Time Frame: Inpatient Day 1, Up to 4 Hours post Session
Population: Pod Users Excluded
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electronic Cigarette | Combustible Cigarette
Number analyzed (Participants) | 33 | 33
score on a scale | 14.4 (6.6) | 14.1 (7.2)

11. Other Pre Specified Outcome: Standardized Session: Half-life
Description: Estimated Time (min) to reduce the plasma nicotine concentration by half based on observed pharmacokinetics.
Time Frame: Inpatient Day 1, Up to 4 Hours post Session
Population: Pod Users Excluded
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Electronic Cigarette | Combustible Cigarette
Number analyzed (Participants) | 33 | 33
min | 137.6 (39.3) | 121.2 (33.9)

ADVERSE EVENTS:
Time Frame: Study participation lasted 2 weeks.
Groups:
- Electronic Cigarette: Electronic cigarette ARM
- Combustible Cigarette: Tobacco Cigarette ARM
Arm/Group | Electronic Cigarette | Combustible Cigarette
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT02470754/Prot_002.pdf
  • Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT02470754/SAP_001.pdf
  • Informed Consent Form (2017-10-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT02470754/ICF_000.pdf